CLINICAL TRIAL: NCT05984719
Title: New Daily Persistent Headache Patient Experience Survey
Brief Title: New Daily Persistent Headache Survey
Acronym: NDPH
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mark J Burish, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-23-0206
Record Dates: First submitted 2023-07-30; First posted 2023-08-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: New Daily Persistent Headache (NDPH); New Daily Persistent Headache
Keywords: Constant headache; Refractory headache disorder
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New daily persistent headache (NDPH) group: Participants with NDPH will be administered an online survey.

SUMMARY:
Purpose: to explore headache characteristics and treatment effects of patient with new daily persistent headache (NDPH) through an online survey.

Research design: Online survey of patients with new daily persistent headache.

Risks: Risks include a breach of confidentiality as well as fatigue from taking the survey online.

Importance of knowledge that may recently be expected to result: The study aims to discover new information in a very understudied disease. This information could, in future studies, help change the diagnostic criteria or lead to new treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NDPH that have been diagnosed by a health care professional (no documentation is needed, participant must simply state that he or she has been diagnosed)

Exclusion Criteria:

* Unable to speak English (the survey is only in English)
* Unable to use a computer to take the online survey

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population is participants with a diagnosis of NDPH. The NDPH diagnosis must come from a physician and will be further assessed with disease-specific survey questions.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Survey data | At study completion, expected to be in 6-12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- UTHealth Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to the online survey - participants can go here directly. (For more information first, call the study team at 713.486.7771 or email the study team at nctt.wec@uth.tmc.edu) — https://redcap.link/ndph